CLINICAL TRIAL: NCT04430816
Title: Management Of Large Incisional Hernia, Double Mesh Modification Of Chevrel's Technique Versus On Lay Mesh Hernioplasty, A Comparative Study
Brief Title: Management Of Large Incisional Hernia, Double Mesh Modification Of Chevrel's Technique Versus On Lay Mesh Hernioplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: compared chevrel hazem
Record Dates: First submitted 2020-06-07; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Hernia Incisional Ventral
Keywords: midline incisional hernia chevrel

STUDY DESIGN:
Intervention Model Description: two groups of patients with incisional hernia group A underwent double mesh modification of chevrel's technique, group B underwent onlay mesh hernioplasty
Who Masked: Participant
Masking Description: the participants don't know the procedure they will undergo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- modified chevrel technique (Active Comparator): 22 participant with large midline incisional hernia underwent repair by double mesh modification of chevrel's technique
  Interventions: Procedure: double mesh modification of chevrel's technique
- ON LAY mesh hernioplasty (Active Comparator): 21 participant with large midline incisional hernia underwent repair by online mesh hernioplasty
  Interventions: Procedure: on lay mesh hernioplasty

INTERVENTIONS:
Procedure: double mesh modification of chevrel's technique — repair of midline incisional hernia by double mesh modification of chevrel's technique
  Arms: modified chevrel technique
Procedure: on lay mesh hernioplasty — repair of midline incisional hernia by online mesh hernioplasty
  Arms: ON LAY mesh hernioplasty

SUMMARY:
comparison between two groups of large midline incisional hernia, the first group managed by double mesh modification of chevrel's technique the second one managed by conventional onlay mesh repair

DETAILED DESCRIPTION:
This comparative study was carried out in general surgery unit, Zagazig university hospitals, between January 2018 and December 2020, on 43 cases with large incisional hernia, participants were randomly allocated according to the deemed option of management into two groups, group A, the modified Chevrel group, 22 participants were treated by double mesh modification of Chevrel's technique, and group B, the on-lay group, participants treated by anatomical repair and fixation of non-absorbable mesh in on-lay position.

inclusion criteria

* > 18 years old suffering large midline incisional hernia. exclusion criteria
* complicated incisional hernia,
* advanced cardiac, respiratory, liver and renal diseases
* patients with abdominal and abdominal wall malignancy
* ASA III and IV The study condition is the large midline incisional hernia defined as hernia following mid line incision, its defect is 10 cm or more in any of its diameters.

The main outcome of the study is recurrence of hernia and local complications mainly skin sloughing, seroma formation and wound infection.

All the study participants signed an informed written consent, the study was approved by our local ethical committee and institutional review board All the study participants were subjected to thorough history taking and full systemic and abdominal examination chest X ray, abdomino-pelvic ultrasound examination, measuring of the defect by ultrasound or abdominal CT if needed, preoperative routine laboratory tests, fractionated heparin was given when indicated as a prophylaxis for deep venous thrombosis (BMI >35, previous history of DVT,), they were given third generation cephalosporins just before the induction of anesthesia.

Procedures :

In participants of the double mesh modification of Chevrel's technique, after excision of the previous scar, skin and subcutaneous tissue was dissected off the hernia sac, the sac was then opened, released off intra-abdominal adhesions and resected, the real defect size was measured, the skin and subcutaneous tissue was dissected off the anterior rectus sheath, dissection was limited to less than 2 cm lateral to the hernia defect edges.

Then, a bilateral vertical incisions of the anterior rectus sheath was done parallel to the midline and at maximum 2 cm far from it thus two medial anterior rectus sheath flaps could be created and dissected off the rectus abdominis muscles on both sides, dissection of both recti abdominis muscles was continued to be separated off the posterior rectus sheath opening the retro-rectus space, linea alba was reformed by suturing each of the newly formed medial anterior rectus sheath flaps to its fellow of the other side, using Vicryl\0 sutures, the flaps help tension free closure of the defect and formation of a common posterior rectus sheath,

A prolene mesh was spread in the retro-rectus space, extending between the two lateral ends of the space and 4 cm beyond the vertical edges of the defect, fixed to the posterior sheath with prolene sutures .

At the end the anterior rectus sheath was closed with prolene mesh tailored to the space between lateral flaps of anterior rectus sheath, and sutured to their medial edges with interrupted non absorbable sutures .

In the group of on-lay mesh repair the old scar was excised, the sac was laid open at its fundus, adhesolysis was done to free the abdominal viscera from the parietal peritoneum, the sac was excised, skin and subcutaneous tissue were dissected of the anterior rectus sheath till the linea semilunaris, taking care to preserve the perforating vessels, anatomical repair was done by midline closure with prolene 1\0 non absorbable interrupted suture, a prolene mesh was fixed in on-lay position by prolene 2\0 sutures.

In both groups after proper hemostasis a suction drain was left over the mesh, subcutaneous tissue was approximated by vicryl 3\0 skin closed by prolene 3\0.in the postoperative period patients received non-steroid pain killer according to need and third generation cephalosporin intravenous injection, wounds were observed after 24 hours for assessment of any local wound complications specially skin flap ischemia, after discharge patients were followed up in the outpatients clinic by the attending surgeon, follow up data including (wound complications as sloughing of skin flap, drainage amount and duration, corset feeling, parasthesia of abdominal wall and corset feeling) was collected in each visit, two months after operation an abdominal wall ultrasound examination was done for detection of early recurrence, a clinic visits or phone contact was done every 6 months till the end of the study.

Continues data was presented in mean and standard deviation, statistically analyzed using t test, z test, in SPSS program 22

ELIGIBILITY:
Inclusion Criteria:

• above 18 years old suffering large midline incisional hernia.

Exclusion Criteria:

* complicated incisional hernia,
* advanced cardiac, respiratory, liver and renal diseases
* patients with abdominal and abdominal wall malignancy
* ASA III and IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of skin flap ischemia | 24 hours postoperative
  impaired capillary filling of wound skin flaps , measured by clinical examination (capillary filling time > 2 seconds)
incidence of seroma formation | 24 hours after drain removal
  presence of more than 20 ml serous fluid collected around the mesh prosthesis measured by superficial probe ultrasound
incidence of hernia recurrence | in the first 2 years post operative
  presence of hernia defect of any size in the midline or near it detected by ultrasound or coputerized tomography scan of the anterior abdominal wall

SECONDARY OUTCOMES:
difference between operative time of both groups | 1 day
  the time between the start point of the operative procedure and the end of the operative procedure

CONTACTS AND LOCATIONS:
Overall Officials: hazem nour, MD, Principal Investigator — zag university
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: No